CLINICAL TRIAL: NCT03108963
Title: L-carnitine Plus Metformin in Clomiphene-resistant Obese PCOS Women, Reproductive and Metabolic Effects: a Randomized Clinical Trial
Brief Title: L-carnitine and Metformin in Obese PCOS Women.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, IBRAHIM ABD ELGAFOR, assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZUH 6
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2017-04

CONDITIONS: PCOS
MeSH Terms: interventions — Carnitine; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-carnitine and Metformin (Experimental): L-carnitine and Metformin in Obese PCOS Women trying induction of ovulation with clomiphene citrate.
  Interventions: Drug: L-carnitine and Metformin
- placebo (Active Comparator): placebo was given toObese PCOS Women trying induction of ovulation with clomiphene citrate.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: L-carnitine and Metformin — L-carnitine plus Metformin was given Obese PCOS Women trying induction of ovulation with clomiphene citrate.
  Other Names: motova plus and glucphage
  Arms: L-carnitine and Metformin
Drug: placebo — placebo was given Obese PCOS Women trying induction of ovulation with clomiphene citrate.
  Arms: placebo

SUMMARY:
L-carnitine and plus metformin in clomiphene-resistant obese PCOS women, reproductive and metabolic effect: a randomized clinical trial

DETAILED DESCRIPTION:
the trial aims to compare L-carnitine and plus metformin in clomiphene-resistant obese PCOS women with placebo to state the reproductive and metabolic effects in form of pregnancy and insulin resistance parameters and lipid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* pco
* obese
* ifertile

Exclusion Criteria:

* no medical disorders
* no hormonal treatment in the previous 3 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 3 momths
  number of women with clinical pregnancy

SECONDARY OUTCOMES:
ovulation rate | 3 momths
  number of women with follicle >18mm.
abortion rate | 3 momths
  number of women with abortions
insulin resistance | 3 momths
  fasting glucose and insulin
lipid metabolism | 3 momths
  Triglyceride, cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim A el sharkwy, MD, Principal Investigator — FACULTY OF MEDICINE ,ZAGAZIG UNIVERSITY
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No